CLINICAL TRIAL: NCT05668078
Title: Evaluating the Effectiveness of an Intervention Involving Rapid Antigen Testing of Students for COVID-19 in Reducing Absences From Schools in Bangladesh
Brief Title: Effectiveness of Rapid Antigen Testing of Students for COVID-19 in Reducing Absences From Schools in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PR-21078
Record Dates: First submitted 2022-11-25; First posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: School Absenteeism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- School-type 1, intervention school-1 (Experimental): We will test all symptomatic students, teachers, and support staff ; and track students symptoms and absenteeism
  Interventions: Diagnostic Test: Rapid Antigen Testing (RAT) for COVID-19
- School-type 2, intervention school-2 (Experimental): We will test all students, teachers, and support staff every 3 days, irrespective of symptoms (also test whenever develops symptoms) and track students symptoms and absenteeism
  Interventions: Diagnostic Test: Rapid Antigen Testing (RAT) for COVID-19
- In School-type 3, control school (Experimental): We will not do any test, only track the students for symptom notification and absenteeism
  Interventions: Diagnostic Test: Rapid Antigen Testing (RAT) for COVID-19

INTERVENTIONS:
Diagnostic Test: Rapid Antigen Testing (RAT) for COVID-19 — COVID-19 RAT intervention done among the school students to see if RAT test can play a role in reducing absenteeism. School type-1-only for symptomatic participants, School type-2-Serial testing at three days interval for all participants and School type-3 got no testing.

SUMMARY:
The goal of this trial is to evaluate the impact of different testing strategies with Rapid Antigen Testing (RAT) on reduction of school absences. RATs are relatively inexpensive, fast, and can be performed at the point of care. Provision of testing in schools will allow rapid identification and isolation of individuals infected with Covid-19. This will likely reduce COVID-19 transmission, as well as allow symptomatic COVID-19 negative students to return to classroom, avoiding the 10-days isolation period. If proven successful, the lessons from this study can be translated to schools in similar settings. While several testing strategies have been proposed and evaluated in developed countries, no studies have evaluated the role of testing for safe operation of schools or reducing absenteeism in developing country contexts.The lessons learned from this study is likely to inform government policy regarding the provision of testing in school.

Study design: Cluster randomized trial

School types: Three types based on testing:

* Intervention school-1: Test all symptomatic students, teachers, and support staff ; and track symptoms and absenteeism
* Intervention school-2: Test all students, teachers, and support staff every 3 days, irrespective of symptoms (also test whenever develops symptoms) and track symptoms and absenteeism
* Control school: Only track the students for symptom notification and absenteeism

DETAILED DESCRIPTION:
Research Design and Methods Study design: Cluster randomized trial School types: Three types based on testing

● School-type 1, intervention school-1: Test all symptomatic participants; and track symptoms and absenteeism

● School-type 2, intervention school-2: Test all participants every three days, irrespective of symptoms (also test whenever develops symptoms), and track symptoms and absenteeism

● In School-type 3, control school: Only track the symptom notification and absenteeism

Trigger testing:

Enrolled students, teachers, and staff will be tested if they are absent from school due COVID-19 like symptoms such as cough, fever, fatigue/ tiredness, headache, loss of taste /loss of smell, sore throat, diarrhoea, shortness of breath/dyspnoea (a person with at least one of the mentioned signs/symptoms at present or within the last five days). These symptoms will be based on the self-report of the individuals. Once a student or staff is absent from school, they will be called to assess their symptoms. If they report COVID-19-like symptoms, they will be asked to come to the testing booth adjacent to their school. If a student arrives at school with any COVID-19-like symptoms or experiences any symptoms during school hours, he/she will be tested immediately.

Study site: Schools in Dhaka, Bangladesh. Selected nine schools

Study Population:

* Students of 9th and 10th grade
* Teachers and support staff Length of data collection: 3 months

Data collection:

Investigator will select three schools meeting the inclusion criteria for the study. Selected schools will be non-residential. The investigator will communicate with the school authorities to confirm their participation prior to the inception of the study. Then invite all the students of classes 9 and 10 and all the teachers and other support staff of the selected school to participate. When the investigator confirms the participant's participation by written consent, collect socio-demographic and health-related information at baseline and begin to follow up with students and teachers.

Sample collection and testing:

Whenever any participant develops any COVID-19-like symptoms, study team will immediately arrange to test their nasal swab samples by Rapid Antigen Test (RAT) on-site and inform them of the result soon after testing. The team will collect two swabs, one for antigen tests and the other for Reverse Transcription Polymerase Chain Reaction (RT-PCR), in case the antigen test is negative. Sample collection to testing completion of RAT may require one hour. Samples that test negative by antigen tests will be tested by RT-PCR, which may take up to 24 hours to get results. Students will stay home until they receive their RT-PCR test results. Swabs will be collected by trained medical technicians of the research team who will be available in school during and after school hours. Sick students will be asked to come to the testing site near the school gate after school hours for testing. The team will collect detailed data on the current signs and symptoms during sample collection. They will also collect information on the current practice of mask use, social distancing, hand washing, travel history, and contact information for the last 14 days from the participants.

Sample testing booth for RAT:

The investigator will select a separate area near the school gate for an on-site sample testing booth. The testing booth area would preferably be inside the school near one side of the school gate, but it can be outside the gate if an arrangement of a booth inside the gate is not suitable. The sample collection booth will remain open after school hours to collect samples who missed school. Two trained medical technologists (MT) of the study team will collect the sample and complete the testing procedure. Both MTs will wear Full PPE during sample collection and ensure standard bio-safety measures while collecting and testing the samples.

If any participants become COVID-19 positive, investigator will recommend ten days of isolation of the positive participant. If the participant is tested negative for RAT and RT-PCR, he/she will continue to attend the school after getting the test result if their health condition permits.

Everyone will be tested routinely in the intervention arm assigned to serial testing, irrespective of their symptoms. In between, if anyone develops symptoms, the team will arrange their sample test immediately.

Communication of test results:

Investigator will send an SMS to the participants immediately with their test results, and positive test results will be communicated via phone and SMS. If anyone needs individual test results, investigator will arrange a hard copy /soft copy of the test report later. Investigator will also send the test results to the school authority by email and or send a hard copy list of test results for their documentation.

RAT testing Kit: "Pnbio COVID-19 AG Papid Tests Device 25T NS".

Outcomes:

1. School absence days due to influenza-like symptoms
2. Episodes of Influenza-like illness (ILI)/COVID-19-like illness Data Analysis Investigator will compare the socio-demographic characteristics between the control and intervention schools using the chi-square test for binary variables and the student's t-test for continuous variables. Each outcome will be undertaken on an 'intention-to-treat (ITT) basis, i.e., all participants with a recorded outcome will be included in the analyses and will be analyzed according to the intervention arm they were allocated. Investigator will model absenteeism rates (number of ill days per student) as a Poisson variable. Investigator will use generalized estimating equations to compare absenteeism rates and COVID-19 incidence between intervention and control schools while accounting for the clustering in the data from each classroom. This comparison will be made in unadjusted and adjusted analyses using multivariate regression models for potential confounders, including SES, family size, health status, mask use, etc

ELIGIBILITY:
Inclusion Criteria:

* A day school (not residential), with at least 50 students per classroom that follows the national curriculum in either Bangla or English instruction
* Students of class Nine, Ten and Eight
* Providing written consent for participation (both student and Guardian)

Exclusion Criteria:

* Not providing written consent for participation (both student and Guardian)

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1141 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
The number of days absent | 10 Weeks
  Daily data on school absence was collected prospectively from the school authorities and the cause of absence was collected from the students.

SECONDARY OUTCOMES:
COVID-19 positivity | 10 Weeks
  Measured from total RAT test done and total RAT positive identified in arm -1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Arifa Nazneen, MBBS, MPH, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No